CLINICAL TRIAL: NCT01293045
Title: Study of Change in Biological Markers of Bone Metabolism Following Consumption of Hydrolyzed Collagen for 3 Months in Healthy, Non-osteoporotic, Menopausal Women.
Brief Title: Biological Bone Markers and Hydrolyzed Collagen Supplement in Menopausal Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nealth Sarl (Network)
Collaborators: ROUSSELOT SAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: ROU_COLHYD09; 2009-A01217-50 (Registry Identifier: AFSSAPS (France))
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2011-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Postmenopausal women; Functional food; Hydrolysed collagen; Bone metabolism; Bone marker of resorption; Bone marker of formation
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HC Group (Experimental): Group of volunteers fed with Hydrolyzed Collagen
  Interventions: Dietary Supplement: hydrolyzed collagen
- CT Group (Active Comparator): Group of volunteers fed with wheat proteins
  Interventions: Dietary Supplement: wheat protein

INTERVENTIONS:
Dietary Supplement: hydrolyzed collagen — 10g/day at breakfast during 90 days
  Arms: HC Group
Dietary Supplement: wheat protein — 10g/day at breakfast during 90 days
  Arms: CT Group

SUMMARY:
* Preliminary scientific studies, in both animals and humans suggest that oral consumption of hydrolyzed collagen acts on the bone remodeling process by stimulating the activity of osteoblasts responsible for bone formation while improving the bone mineral density and biomechanical resistance of long bones.
* The objective of this clinical research is to measure changes in biomarkers of bone turnover in postmenopausal healthy women, not osteoporotic, in response to consumption of hydrolyzed collagen for three months.
* For this, we propose to measure blood and urinary markers of formation and bone resorption before consumption, then 45 and 90 days after daily consumption of 10 g of hydrolyzed collagen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Aged between 55 and 65 years
* Primary or secondary amenorrhea for at least 5 years
* BMI ≥ 20 kg/m2 and < 27 kg/m2
* DXA > 2.5 SD
* No history of fragility fracture bone
* Not under guardianship
* Not on hormone replacement or any osteoporotic therapy
* Covered by Social Security
* Negative serology for hepatitis B/C and HIV
* Written informed consent form signed.

Exclusion Criteria:

* Bone density < 2.5 SD (standard deviation)
* Endocrine disease
* No history of fragility fracture bone
* Dietary disorder (anorexia, bulimia)
* Hormone replacement therapy
* Inclusion in another clinical study
* Subjects receiving over 4,500 Euros in the last 12 months (including the present study)
* Subjects presenting risk of non-compliance in the opinion of the recruiting doctor.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Serum C-terminal telopeptide of type 1 collagen (CTX) | Day 45
  MARKERS OF BONE RESORPTION : change from Baseline (Day 0) in serum CTX at 45 days

SECONDARY OUTCOMES:
Urinary telopeptide N-terminal of type 1 collagen (NTX) | Day 45
  MARKERS OF BONE RESORPTION : change from Baseline (Day 0) in urinary NTX at 45 days
Serum osteocalcin | Day 45
  MARKERS OF BONE FORMATION : change from Baseline (Day 0) in serum osteocalcin at 45 days
Serum bone alkaline phosphatase | Day 45
  MARKERS OF BONE FORMATION: change from Baseline (Day 0) in serum bone alkaline phosphatase at 45 days
Serum amino-terminal pro-peptide of type 1 procollagen (P1NP) | Day 45
  MARKERS OF BONE FORMATION : change from Baseline (Day 0) in serum P1NP at 45 days
Urinary telopeptide N-terminal of type 1 collagen (NTX) | Day 90
  MARKERS OF BONE RESORPTION : change from Baseline (Day 0) in urinary NTX at 90 days
Serum osteocalcin | Day 90
  MARKERS OF BONE FORMATION : change from Baseline (Day 0) in serum osteocalcin at 90 days
Serum bone alkaline phosphatase | Day 90
  MARKERS OF BONE FORMATION: change from Baseline (Day 0) in serum bone alkaline phosphatase at 90 days
Serum amino-terminal pro-peptide of type 1 procollagen (P1NP) | Day 90
  MARKERS OF BONE FORMATION : change from Baseline (Day 0) in serum P1NP at 90 days
Serum C-terminal telopeptide of type 1 collagen (CTX) | Day 90
  MARKERS OF BONE RESORPTION : change from Baseline (Day 0) in serum CTX at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert BENAMOUZIG, MD, PhD, Principal Investigator — Centre de Recherche en Nutrition Humaine d'Ile-de-France
Locations (1):
- CRNH - Centre de Recherche sur Volontaires - Hôpital AVICENNE, Bobigny, Seine-saint-denis, France

REFERENCES:
- [Background] Nomura Y, Oohashi K, Watanabe M, Kasugai S. Increase in bone mineral density through oral administration of shark gelatin to ovariectomized rats. Nutrition. 2005 Nov-Dec;21(11-12):1120-6. doi: 10.1016/j.nut.2005.03.007. PMID 16308135
- [Background] Takeuchi Y, Nakayama K, Matsumoto T. Differentiation and cell surface expression of transforming growth factor-beta receptors are regulated by interaction with matrix collagen in murine osteoblastic cells. J Biol Chem. 1996 Feb 16;271(7):3938-44. doi: 10.1074/jbc.271.7.3938. PMID 8632016
- [Background] Wu J, Fujioka M, Sugimoto K, Mu G, Ishimi Y. Assessment of effectiveness of oral administration of collagen peptide on bone metabolism in growing and mature rats. J Bone Miner Metab. 2004;22(6):547-53. doi: 10.1007/s00774-004-0522-2. PMID 15490264
- [Background] Guillerminet F, Beaupied H, Fabien-Soule V, Tome D, Benhamou CL, Roux C, Blais A. Hydrolyzed collagen improves bone metabolism and biomechanical parameters in ovariectomized mice: an in vitro and in vivo study. Bone. 2010 Mar;46(3):827-34. doi: 10.1016/j.bone.2009.10.035. Epub 2009 Nov 4. PMID 19895915